CLINICAL TRIAL: NCT02700139
Title: Shamir Aspheric Ophthalmic Lenses (MyLens) for Myopic Control Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A corporate decision to terminate the study
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Shamir Optical Industry Ltd (Industry)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20160105001
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Myopia
Keywords: Myopia control, aspheric lenses, children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspheric lens (Experimental): An aspheric lens which is supposed to slow myopic progression in children by unique asphericity (proprietary information)
  Interventions: Device: Aspheric lens
- Single vision spheric/toric lenses (No Intervention): Control: single vision spheric/toric lenses

INTERVENTIONS:
Device: Aspheric lens — By using a special asphericity, MyLens is customized for various prescriptions and vision directions based on specific measurements, intended for myopia correction and control
  Other Names: MyLens
  Arms: Aspheric lens

SUMMARY:
The aim of this clinical trial is to compare the rate of myopic progression in children wearing aspheric (MyLens) and spherical/ toric ophthalmic lenses. The proposed lens design is an aspheric lens which is supposed to slow myopic progression in children by unique asphericity (proprietary information). Myopic progression is quantified by changes in axial length (AL) and cycloplegic refractive error (Rx) will be monitored for 6-12 months (6 months crossover) with double-masking. Peripheral refraction and ocular aberration will be evaluated.

DETAILED DESCRIPTION:
Visual manipulation induced by progressive addition lenses (PALs) have been shown to inhibit eye growth and myopia development in children with up to 11% to 21% efficacy compared to single vision lenses. However, the treatment effect of PALs is statistically significant but clinically insufficient. The current study aims at investigating the use of spectacle lenses with a unique novel design for myopia control in children. This prospective one-year randomized clinical study will evaluate axial elongation and myopia progression in eyes using the novel lens design compared to those using the conventional single-vision design. It is a double-masked, cross-over study. One eye will be fitted with the study lens and the other eye will be fitted with the single-vision lens. Subjects will be asked to wear the spectacles for 6 months and the two lens designs will be swapped in the next 6 months after a wash-out period of 2 weeks. Both the subjects and examiners will not aware the lens design being used by the subjects in each phase.

ELIGIBILITY:
Inclusion Criteria:

* Myopia between 0.75 ~ - 4.50 D and with-the-rule astigmatism not more than 1.50 D
* Difference between eyes, no more than 1.25 spherical equivalent
* Best corrected visual acuity (VA) is equal to or better than 0.10 in logMAR scale (Snellen VA 6/7.5 or better)
* Eyes straight at distance and near with best subjective correction
* Willing to be randomized and wear the study spectacles according to the instructions from practitioner
* Willing to come back for follow up in the Optometry Clinic during the study period

Exclusion Criteria:

* Abnormal ocular and general health
* Prior myopic treatment (e.g. refractive surgery and progressive lens wear for myopic control) before and during the study period
* History of rigid contact lenses (including orthokeratology lenses) wearing
* Systemic condition which might affect refractive development (for example, Down syndrome, Marfan's syndrome)
* Ocular conditions which might affect the refractive error (for example, cataract, ptosis).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changes in axial length in 6-12 months | Every 6 months for a period of 1 year
  Evaluate the changes in cycloplegic axial length in the eye with aspheric lens (MyLens) compared to the other eye with single vision spheric/toric lens

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The demographic data of subjects recruited in this study will be disclosed in this website

REFERENCES:
- [Background] Edwards MH, Li RW, Lam CS, Lew JK, Yu BS. The Hong Kong progressive lens myopia control study: study design and main findings. Invest Ophthalmol Vis Sci. 2002 Sep;43(9):2852-8. PMID 12202502
- [Background] Gwiazda J, Hyman L, Hussein M, Everett D, Norton TT, Kurtz D, Leske MC, Manny R, Marsh-Tootle W, Scheiman M. A randomized clinical trial of progressive addition lenses versus single vision lenses on the progression of myopia in children. Invest Ophthalmol Vis Sci. 2003 Apr;44(4):1492-500. doi: 10.1167/iovs.02-0816. PMID 12657584
- [Background] Hasebe S, Jun J, Varnas SR. Myopia control with positively aspherized progressive addition lenses: a 2-year, multicenter, randomized, controlled trial. Invest Ophthalmol Vis Sci. 2014 Sep 30;55(11):7177-88. doi: 10.1167/iovs.12-11462. PMID 25270192
- [Background] Hasebe S, Ohtsuki H, Nonaka T, Nakatsuka C, Miyata M, Hamasaki I, Kimura S. Effect of progressive addition lenses on myopia progression in Japanese children: a prospective, randomized, double-masked, crossover trial. Invest Ophthalmol Vis Sci. 2008 Jul;49(7):2781-9. doi: 10.1167/iovs.07-0385. PMID 18579755
- [Background] Yang Z, Lan W, Ge J, Liu W, Chen X, Chen L, Yu M. The effectiveness of progressive addition lenses on the progression of myopia in Chinese children. Ophthalmic Physiol Opt. 2009 Jan;29(1):41-8. doi: 10.1111/j.1475-1313.2008.00608.x. PMID 19154279